CLINICAL TRIAL: NCT04122677
Title: Performance and Safety of the Polylactic Interference Screw Used in Anterior Cruciate Ligament Reconstructions
Status: Completed | Type: Observational
Sponsor: Biomatlante (Industry)
Collaborators: Atlanstat (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-A03207-48
Record Dates: First submitted 2019-09-30; First posted 2019-10-10 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Knee Ligament Injury
Keywords: Knee Ligament Injury; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Reconstruction; Knee Ligament Rupture; Knee Ligament Reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Anterior Cruciate Ligament Reconstruction — Reconstruction of the Anterior Cruciate Ligament using an interference screw.

SUMMARY:
The evaluation of the clinical data has demonstrated the conformity of the Polylactic Interference Screw (PIS), with the relevant essential requirements for its use in orthopaedic applications. The Polylactic Interference Screws are intended for tibial and femoral ligament/graft fixation in the case or Anterior Cruciate Ligament (ACL) reconstructions. It has been concluded that the risks associated with the use of the device are acceptable when weighted against the benefits to the patients. In order to improve the clinical data on the PIS, the manufacturer, Biomatlante, decided to assess that the performance and safety of the device are maintained until the reaching of its intended use. In this objective, the goal of this study will be to observe the following parameters:

Objective IKDC score (clinical evaluation) Subjective IKDS score (functional evaluation) Safety (report of any adverse event) Follow-up of the patient's recovery

ELIGIBILITY:
Inclusion Criteria:

* Acute or chronic Anterior Cruciate Ligament deficiency with complete or partial lesion of the anteromedial bundle requiring primary reconstruction of the Anterior Cruciate Ligament with hamstring tendons
* Males or females aged from 18 to 60 years
* No history of surgery on the affected knee
* Patients not under guardianship or judicial protection
* Signature of non opposition form (consent of the patient

Exclusion Criteria:

* History of ligament, meniscal surgery or fracture of the affected knee
* Pregnancy of breastfeeding women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population is considered as all the patients included in the study that meet the inclusion and exclusion criteria.
  The study population is composed of 56 patients according to the protocol.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Change of the objective International Knee Documentation Committee score before and after surgery | 4 months before surgery / 7 months post-surgery
  Record of the objective International Knee Documentation Committee score (A = normal, B = almost normal, C = abnormal or D = very abnormal)
Change of the subjective International Knee Documentation Committee score before and after surgery | 4 months before surgery / 7 months post-surgery
  Record of the subjective International Knee Documentation Committee score (from 1 to 100 where 100 is the best result)

SECONDARY OUTCOMES:
Number and precise description of any adverse event during the follow-up | Before surgery until 7 months post-surgery
  Record and description of any adverse event during the follow-up that reflects the safety of the Polylactic Interference Screw
Change in the patients recovery | 2 months post-surgery
  Record of specific items of the Objective International Knee Documentation Committee score reflecting the patients recovery

CONTACTS AND LOCATIONS:
Overall Officials: François-Xavier FV VERDOT, M.D., Principal Investigator — Centre ORTHEO
Locations (1):
- Centre ORTHEO, Saint-Étienne-de-Montluc, Pays de la Loire Region, France

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-07-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT04122677/Prot_000.pdf